CLINICAL TRIAL: NCT01536054
Title: A Phase I Clinical Trial of mTOR Inhibition With Sirolimus for Enhancing ALVAC(2)-NY-ESO-1(M)/TRICOM Vaccine Induced Anti-Tumor Immunity in Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Sirolimus and Vaccine Therapy in Treating Patients With Stage II-IV Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 199911; NCI-2011-02964 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-30; First posted 2012-02-20 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Epithelial Cancer; Stage IIA Primary Peritoneal Cavity Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Epithelial Cancer; Stage IIB Primary Peritoneal Cavity Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Epithelial Cancer; Stage IIC Primary Peritoneal Cavity Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Primary Peritoneal Cavity Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Sirolimus; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vaccine, sirolimus, GM-CSF) (Experimental): Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine SC on day 1 and GM-CSF SC on days 1-4. Patients also receive sirolimus PO QD on days 1-14 OR 15-28 OR 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive an additional course of ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine only followed by ALVAC(2)-NY-ESO-I (M)/TRICOM vaccine SC 8 weeks after completion of course 4.
  Interventions: Biological: ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine; Drug: sirolimus; Other: laboratory biomarker analysis; Biological: sargramostim

INTERVENTIONS:
Biological: ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine — Given SC
  Other Names: vCP2292
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Other: laboratory biomarker analysis — Correlative studies
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine

SUMMARY:
This phase I trial studies the side effects and best dose and schedule of sirolimus when given together with vaccine therapy in treating patients with stage II-IV ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer. Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy together with sirolimus may be an effective treatment for ovarian, fallopian tube, or primary peritoneal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine with sirolimus at varying dose and schedule.

SECONDARY OBJECTIVES:

I. To determine the effectiveness of sirolimus on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity: peripheral blood NY-ESO-1 specific cluster of differentiation (CD)8+ and CD4+ T-cells; peripheral blood NY-ESO-1 specific antibodies; peripheral blood frequency of CD4+CD25+forkhead box P3 (FOXP3)+ regulatory T-cells.

II. Explore time to disease progression.

OUTLINE: This is a dose-escalation study of sirolimus.

Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine subcutaneously (SC) on day 1 and sargramostim (GM-CSF) SC on days 1-4. Patients also receive sirolimus orally (PO) once daily (QD) on days 1-14 OR 15-28 OR 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive an additional course of ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine only followed by ALVAC(2)-NY-ESO-I (M)/TRICOM vaccine SC 8 weeks after completion of course 4.

After completion of study treatment, patients are followed up at 30 days, and 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be women with stages II-IV epithelial ovarian, fallopian tube, or primary peritoneal carcinoma who have completed standard therapy for primary or recurrent disease (i.e., patients who would normally be observed); eligible patients may have asymptomatic residual measurable disease on physical examination and/or computed tomography (CT) scan, and/or may have an elevated cancer antigen 125 (CA-125); or may be in complete clinical remission after treatment for primary or recurrent disease; these patients would normally enter a period of observation after standard management
* Any human leukocyte antigen (HLA) type; (historic HLA typing is permitted)
* Tumor expression of NY-ESO-1 or cancer/testis antigen 2 (LAGE-1) by immunohistochemistry (IHC) and/or real-time polymerase chain reaction (RT-PCR)
* No allergy to eggs
* Life expectancy > 6 months
* Hematology and biochemistry laboratory results within the limits normally expected for the patient population, without evidence of major organ failure
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelet >= 75,000/uL
* Hemoglobin (Hgb) >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) =< 3 x ULN
* Serum creatinine =< 2 x ULN
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5
* Electrocardiogram, showing no evidence of congestive heart failure, myocardial infarction, and cardiomyopathy
* Have been informed of other treatment options
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 2
* Demonstrate the ability to swallow and retain oral medication
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patients may have received previous NY-ESO-1 vaccine therapy

Exclusion Criteria:

* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g. serious infections requiring antibiotics, bleeding disorders)
* History of severe autoimmune disorders requiring use of steroids or other immunosuppressives
* Concomitant systemic treatment with corticosteroids, anti-histamine or nonsteroidal anti-inflammatory drugs and other platelet inhibitory agents, strong inhibitors/inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP450-3A4)
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study drug (6 weeks for nitrosoureas); concomitant hormonal therapies for breast cancers are allowed
* Known allergy or history of life threatening reaction to GM-CSF
* Clinically significant heart disease (N-YHA Class III or IV)
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study drug
* Known hepatitis B, hepatitis C, or HIV
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Known pulmonary hypertension
* Known hypersensitivity to sirolimus
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug; (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk by participating in this study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2015-04-21 (Actual); Study Completion 2015-04-21 (Actual)

PRIMARY OUTCOMES:
Safety of ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine in combination with varying dose levels and schedules of sirolimus, assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 30 days after completion of study treatment
  The toxicity rate will be estimated using a one-sided, 95%, exact binomial confidence interval (Clopper-Pearson). The lower one sided limit will be used.

SECONDARY OUTCOMES:
Effectiveness of sirolimus on enhancing vaccine efficacy, assessed by NY-ESO-1 specific cellular and humoral immunity | Up to 1 year
  The following parameters will be determined: (I) generation of memory T-cells with (2) high avidity that are also (3) resistant to regulatory T cells (Tregs): (4) secondary recall responses. Analyzed via an analysis-of-covariance (ANCOVA) model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design. The biological signal across all cohorts will be tested on whether or not the slope parameter is 0 or not.
Antibody titers | At baseline, days 29, 57, 85, 141, and at 6 weeks-post treatment
  Will be analyzed via an ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design.
NY-ESO-1 specific CD8+ and CD4+ frequency and function | At baseline, days 1, 29, 57, 85, 113, 141, and at 6 weeks-post treatment
  The analysis of continuous immunological response endpoints will be analyzed via an ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design.
Frequency of memory T-cell populations | At baseline, days 1, 29, 57, 85, 113, 141, and at 6 weeks-post treatment
  The analysis of continuous immunological response endpoints will be analyzed via an ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design.
TCR avidity | At baseline, days 1, 29, 57, 85, 113, 141, and at 6 weeks-post treatment
  The analysis of continuous immunological response endpoints will be analyzed via an ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design.
Secondary recall response | Up to 1 year
  The analysis of continuous immunological response endpoints will be analyzed via an ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 x 3 design.
Time to disease progression | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Background] Odunsi K, Matsuzaki J, James SR, Mhawech-Fauceglia P, Tsuji T, Miller A, Zhang W, Akers SN, Griffiths EA, Miliotto A, Beck A, Batt CA, Ritter G, Lele S, Gnjatic S, Karpf AR. Epigenetic potentiation of NY-ESO-1 vaccine therapy in human ovarian cancer. Cancer Immunol Res. 2014 Jan;2(1):37-49. doi: 10.1158/2326-6066.CIR-13-0126. PMID 24535937
- [Background] Liao J, Qian F, Tchabo N, Mhawech-Fauceglia P, Beck A, Qian Z, Wang X, Huss WJ, Lele SB, Morrison CD, Odunsi K. Ovarian cancer spheroid cells with stem cell-like properties contribute to tumor generation, metastasis and chemotherapy resistance through hypoxia-resistant metabolism. PLoS One. 2014 Jan 7;9(1):e84941. doi: 10.1371/journal.pone.0084941. eCollection 2014. PMID 24409314
- [Background] Godoy HE, Khan AN, Vethanayagam RR, Grimm MJ, Singel KL, Kolomeyevskaya N, Sexton KJ, Parameswaran A, Abrams SI, Odunsi K, Segal BH. Myeloid-derived suppressor cells modulate immune responses independently of NADPH oxidase in the ovarian tumor microenvironment in mice. PLoS One. 2013 Jul 26;8(7):e69631. doi: 10.1371/journal.pone.0069631. Print 2013. PMID 23922763
- [Background] Matsuzaki J, Tsuji T, Luescher I, Old LJ, Shrikant P, Gnjatic S, Odunsi K. Nonclassical antigen-processing pathways are required for MHC class II-restricted direct tumor recognition by NY-ESO-1-specific CD4(+) T cells. Cancer Immunol Res. 2014 Apr;2(4):341-50. doi: 10.1158/2326-6066.CIR-13-0138. Epub 2013 Dec 17. PMID 24764581
- [Derived] Withers HG, Matsuzaki J, Long M, Rosario SR, Chodon T, Tsuji T, Koya R, Yan L, Wang J, Keler T, Lele SB, Zsiros E, Lugade A, Hutson A, Blank S, Bhardwaj N, Shrikant P, Liu S, Odunsi K. mTOR inhibition modulates vaccine-induced immune responses to generate memory T cells in patients with solid tumors. J Immunother Cancer. 2025 Mar 25;13(3):e010408. doi: 10.1136/jitc-2024-010408. PMID 40132910